CLINICAL TRIAL: NCT02816788
Title: Investigation of Equine Assisted Therapy for Post-Traumatic Stress Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Variety of issues, including imminent retirement of principal investigator.
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Anne Barnfield, Dr., Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108102
Record Dates: First submitted 2016-06-16; First posted 2016-06-29 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Equine Assisted Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Single group, within subjects comparison. Pre- and post-intervention comparisons.
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Equine Assisted Therapy (EAT) (Experimental): Equine Assisted Therapy (EAT) treatment group
  Interventions: Behavioral: Equine Assisted Therapy (EAT)

INTERVENTIONS:
Behavioral: Equine Assisted Therapy (EAT) — Psychotherapy incorporating use of equines (Equine Assisted Therapy; EAT) to facilitate therapy to improve the social, emotional and psychological well-being of participants and alleviate PTSD symptoms.

SUMMARY:
In partnership with SARI Therapeutic Riding (SARI TR) and other equine therapy locations, Brescia University College, at the University of Western Ontario, will study the use of Equine Assisted Therapy (EAT) for military veterans and "first reponders" (emergency services personell) diagnosed with Post-Traumatic Stress Disorder. Data will be collected through tests and questionnaires, and follow-up interviews with participants. It is expected that after a series of EAT sessions, the social, emotional and psychological well-being of participants will be improved and PTSD symptoms alleviated.

DETAILED DESCRIPTION:
The objective of this study is to evaluate outcomes of participation in Equine Assisted Therapy for those with a history of PTSD.

This study protocol will be a within subjects design: Treatment group with pre- and post-intervention comparisons. Participants will be Military Veterans and "first responders" (emergency services personell) with prior diagnosis of PTSD; N=8 to 10.

Procedures for treatment group: The treatment group will engage in sets of EAT sessions to be run at SARI Therapeutic Riding (SARI TR) and other equine therapy locations. A typical EAT session will involve beginning the session by checking in as a group, engaging in one or two activities with the horses and then processing the activity as a group. Each session will also end with a check out. The activities with equines will range from observation/educational, grooming, reflective work involving creative expression with writing/art, or more active activities such as leading. Each session will have an overall topic which will provide the framework for the session. Interactions with equines will take place in the indoor arena (an enclosed space for riding/training horses), whilst other aspects of the sessions will take place in the main lounge. Sessions will be conducted by a Clinical Counsellor certified with their Provincial Counselling and Psychotherapy Association, assisted by other certified personnel, including those with horse handling experience. Each session will include up to eight to ten participants. There will be two persons with therapeutic expertise and one with horse/TR experience attending to participants at all times during interaction with equines. Sessions will usually last about two and a half hours, incorporating psychotherapy and interacting with equines, over a course of several sessions.

General procedure: Military Veterans and first responders with PTSD will be recruited from the local Occupational Stress Injury Social Support (OSISS) PTSD support group and similar organizations. This service "is a partnership program between the Department of National Defence and Veterans Affairs Canada" (OSISS website) created to provide peer support to Canadian Forces personnel, Veterans and their families. The OSISS provides peer support and aids in linking members to appropriate services, programmes and supports. Data will be collected through questionnaire-type tests and post-session interview of participants. A set of short tests, the Rosenberg Self-esteem Scale, the Positive and Negative Affect Scale (PNAS), and the PTSD Checklist for DSM-5 (PCL-5) will be administered. Participants will complete sets of tests at pre-session, post-session, and follow-up, and will be interviewed one week after the end of the study in order to obtain further data. Longer-term follow-up is also anticipated, with measures being repeated at further time points (e.g., one-, three-, and six-month follow-up) after completion of EAT sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Post-Traumatic Stress Disorder (PTSD)
* with veteran or "first responder" status
* Both of these ascertained by self-report, confirmed by membership in Occupational Stress Injury Social Support (OSISS) group or similar organization

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Understanding of effects/effectiveness of EAT for PTSD. | 6 months
  PTSD Checklist for Diagnostic and Statistical Manual-5 (PCL-5)

SECONDARY OUTCOMES:
Understanding of effects/effectiveness of EAT for PTSD-related moods and emotions. | 6 months
  Positive and Negative Affect Scale (PNAS)
Understanding of effects/effectiveness of EAT for PTSD-related self esteem issues. | 6 months
  Rosenberg Self Esteem Scale

CONTACTS AND LOCATIONS:
Overall Officials: Anne MC Barnfield, PhD, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duncan, R., Critchley, S., & Marland, J. (2014). Can Praxis: A Model of Equine Assisted Learning (EAL) for PTSD. Canadian Military Journal 14(2), 64-69.
- [Background] Johnson, R. A. (2015). Effects of Equine Assisted Activities on PTSD Symptoms, Coping Self-Efficacy, Emotion Regulation, and Social Engagement in Military Veterans. Horses and Humans Research Foundation Final Grant Reporting. Retrieved from: http://www.horsesandhumans.org/RA_Johnson_Final_Grant_Report_12-2015.pdf
- [Background] Yorke, J., Adams, C., &Coady, N. (2008). Therapeutic value of equine-human bonding in recovery from trauma. Anthrozoös, 21(1), 17-33.
- [Background] Barnfield, A. M. C. (2015). A response to Anestis, Anestis, Zawilinski, Hopkins and Lilienfeld (2014). Scientific and Educational Journal of Therapeutic Horse Riding, 2015, 10-15.